CLINICAL TRIAL: NCT05725174
Title: Volatile Non-Invasive Biomarkers of Epileptic Seizures
Acronym: VIBES
Status: Recruiting | Type: Observational
Sponsor: University College London Hospitals (Other)
Collaborators: Imperial College London (Other)
Responsible Party: Principal Investigator, Eleonora Lugara, Dr, University College London Hospitals
Other Study IDs: 285913; 22/LO/0808 (Other: REC Reference)
Record Dates: First submitted 2023-02-02; First posted 2023-02-13 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Epilepsy; Non-Epileptic Seizure
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Sample Collection — Patients will have breath samples collected by blowing into a bag, and sweat samples collected by gauze. These samples will be collected at various timepoints whilst the patients are admitted on the ward.

SUMMARY:
Breath and sweat samples will be collected from people who have been admitted to hospital after a potential seizure and analysed by the team. The researchers then hope to identify a pattern of small molecules that can distinguish seizures from other events, and perhaps determine the severity of the seizure.

DETAILED DESCRIPTION:
Determining whether someone has had an epileptic seizure, or another event, can be challenging and result in the wrong diagnosis. A 'seizure test' used after the event would therefore be very helpful.

Researchers have used small molecules released from the body in breath and sweat to detect cancers and other diseases; this study will determine whether a similar method can be used to detect whether someone has had an epileptic seizure.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have been admitted to either University College London's Queen's Square EEG-telemetry unit or Chalfont Centre for Epilepsy, for diagnosis of seizure events.
2. Patients aged 18 years or above

Exclusion Criteria:

1. Patients with active infection or who have taken antibiotics within 4 weeks
2. Patients on immunosuppressive medications
3. Patients with co-morbidities preventing breath collection
4. Patients unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with a diagnosis of epileptic or non-epileptic seizures
Sampling Method: Non-Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Distinguishing epileptic from non-epileptic seizures | 3 years
  To distinguish epileptic from non-epileptic seizures with the detection of volatile organic compounds (VOCs) in breath and sebum samples.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Walker, MB BChir FRCP, Principal Investigator — Professor
Locations (2):
- United Kingdom (2):
  - Chalfont Centre for Epilepsy, London, Buckinghamshire
  - National Hospital for Neurology and Neurosurgery, London, London

IPD SHARING:
Plan to Share IPD: Undecided
If necessary, anonymised data will be shared with other researchers in a case by case scenario. For anonymised data to be shared with commercial entities, a research contract will need to be evaluated.